CLINICAL TRIAL: NCT03126318
Title: A Phase 1 Randomized, Double-Blind, Placebo-Controlled, Cohort Dose-Escalation Study in Patients With Chronic Kidney Disease to Assess the Safety, Pharmacokinetics, and Pharmacodynamics of a Single Dose of COR-001 (COR-001-SC1)
Brief Title: A Study of Patients With Chronic Kidney Disease to Assess the Safety of a Single Dose of COR-001
Acronym: COR-001-SC1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Corvidia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16-2272
Record Dates: First submitted 2017-04-05; First posted 2017-04-24 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo-controlled - 4 cohorts of 4 patients each with a dosing regimen of 3:1 (active:placebo)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- COR-001 (Active Comparator): COR-001 5, 15, 50, or 100 mg dose (depending on dose cohort assigned to patient) given by subcutaneous injection one time only
  Interventions: Drug: COR-001
- Placebo (Placebo Comparator): Placebo at pH 6.0will be given in a volume to match the volume of COR-001 being given for the dose cohort by subcutaneous injection one time only
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: COR-001 — Anti-inflammatory therapy
  Arms: COR-001
Drug: Placebo — Sterile water with a final buffer of 25 mM Histidine, 8.5% (w/v) trehalose and 0.05% PS80
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled trial designed to evaluate the safety, pharmacokinetics, and pharmacodynamic effects of a single dose of the study drug or placebo administered subcutaneously to patients with moderate-to-severe chronic kidney disease and persistent inflammation.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled trial designed to evaluate the safety, pharmacokinetics, and pharmacodynamic effects of a single dose of the study drug or placebo administered subcutaneously to patients with moderate-to-severe chronic kidney disease (CKD) and persistent inflammation (defined as a persistently elevated serum CRP (C-Reactive Protein) level). The primary objective is to evaluate the safety of a single dose of the study drug delivered subcutaneously. Four CKD patients will be randomized to the study drug or placebo within each dosing cohort in a ratio of 3:1. The dosing cohorts are 5 mg, 15 mg, 50 mg, and 100 mg. Each patient will be given 1 dose of the study drug and then be followed for 12 weeks for primary safety, pharmacokinetic and pharmacodynamic assessments. Next, patients will continue to be followed for an additional 20 weeks (32 weeks observation in total) for safety and anti-drug antibody assessments.

Prior to dose escalation (i.e., higher total dose than studied in the preceding cohorts), there will be a formal safety review and the data will have been determined to be acceptable by a Data Safety Monitoring Board (DSMB) which will include at least one nephrologist. The safety review required for dose escalation will include at least 21 days of treatment data from the preceding cohort(s). The DSMB will also meet to review data concerning an SAE (Serious Adverse Event) that is suspected to be study drug related

The investigative team (other than an un-blinded research pharmacist or equivalent) will be blinded to the treatment assignment.

ELIGIBILITY:
Inclusion Criteria:

1. CKD stage III or IV
2. Serum CRP > 2 mg/L measured twice during the Screening period at least one week apart
3. Urine protein excretion < 3.5 g/24h estimated by a spot urine protein/creatinine ratio
4. The patient agrees to comply with the contraception and reproduction restrictions of the study - use 2 forms of acceptable contraception

Exclusion Criteria:

1. Patients with advanced CKD requiring chronic dialysis
2. Hospitalization over the period of 6 weeks prior to randomization
3. Use of systemic immunosuppressive drugs during the Screening Period or anticipated use of such drugs anytime during the study Note: Use of otic, ophthalmic, inhaled, and topical corticosteroids or local corticosteroid injections are not exclusionary.
4. History of or expected to undergo living related kidney transplant during the study period
5. Currently receiving or planning to receive live or inactivated vaccines
6. Clinical evidence or suspicion of active or smoldering infection (e.g., diabetic foot ulcer) or use of antibiotics during the Screening period
7. History of a positive PPD or prior diagnosis of tuberculosis
8. Evidence of HIV infection or carrier state by serology at Screening
9. Hepatitis B or C by serology (i.e. Hepatitis B Surface Antigen or Hepatitis C antibody positive) at Screening
10. AST or ALT > 2.5x ULN at Screening
11. History of liver cirrhosis or home oxygen use
12. History of gastrointestinal ulceration or active diverticulitis in the 1 year prior to Screening
13. Absolute neutrophil count < 2 x 109/L at Screening
14. Platelet count < 100 x 109/L at Screening
15. Participated in an investigational drug study within 30 days of Screening or Screening is within 5 half-lives of the investigational compound.
16. Known allergy to the study drug or any of its ingredients
17. Breastfeeding or a positive pregnancy test at Screening or Day -1.
18. Any condition that could interfere with, or for which the treatment might interfere with, the conduct of the study or interpretation of the study results, or that would in the opinion of the Investigator increase the risk of the subject's participation in the study.

    This would include but is not limited to alcoholism, drug dependency or abuse, psychiatric disease, epilepsy, anemia attributable to a primary hematologic disease (e.g., sickle cell anemia), or any unexplained blackouts.
19. Actively treated malignancy (other than non-melanoma skin cancers) during the 1 year prior to Screening. Patients receiving hormonal treatment only during this period only may be enrolled with the approval of the medical monitor.
20. Myocardial infarction during the 3 months prior to Screening or during Screening
21. Severe arthritis, lupus, inflammatory bowel disease, asthma or other disease(s) or medical condition(s) that, in the opinion of the investigator, could interfere with hs-CRP or immune function
22. Use of CYP substrates with a narrow therapeutic index (please see detailed table below).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-05-19 (Actual); Primary Completion 2019-03-14 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
The safety of a 5 mg dose of COR-001 as measured by the incidence of adverse events | 1 month after the 4th patient has received study drug
  To evaluate the safety of a 5 mg dose of COR-001 delivered subcutaneously
The safety of a 15 mg dose of COR-001 as measured by the incidence of adverse events | 1 month after the 4th patient has received study drug
  To evaluate the safety of a 15 mg dose of COR-001 delivered subcutaneously
The safety of a 50 mg dose of COR-001 as measured by the incidence of adverse events | 1 month after the 4th patient has received study drug
  To evaluate the safety of a 50 mg dose of COR-001 delivered subcutaneously
The safety of a 100 mg dose of COR-001 as measured by the incidence of adverse events | 1 month after the 4th patient has received study drug
  To evaluate the safety of a 100 mg dose of COR-001 delivered subcutaneously

SECONDARY OUTCOMES:
Pharmacokinetic analysis: maximum serum drug concentrations (Cmax) | Pre-dose, 4 hours post-dose, and days 2-7, 11, 15, 22, 29, 57, 85, 141, and 225 post-dose.
  To evaluate single-dose pharmacokinetics of COR-001 delivered subcutaneously
Pharmacokinetic analysis: area under the serum drug concentration-time curve (AUC) | Pre-dose, 4 hours post-dose, and days 2-7, 11, 15, 22, 29, 57, 85, 141, and 225 post-dose.
  To evaluate the single-dose pharmacokinetics of COR-001 delivered subcutaneously
Pharmacokinetic analysis: terminal elimination half-life (t1/2) | Pre-dose, 4 hours post-dose, and days 2-7, 11, 15, 22, 29, 57, 85, 141, and 225 post-dose.
  To evaluate the single-dose pharmacokinetics of COR-001 delivered subcutaneously
The effectiveness of COR-001 as measured by levels of an inflammatory marker | Screening and at weeks 1 - 5, 8, 12, 20, and 32.
  To evaluate the effectiveness of COR-001 as measured by CRP levels.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Chonchol, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Coloardo Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nowak KL, Kakkar R, Devalaraja M, Lo L, Park W, Gobburu J, Kling D, Davidson M, Chonchol M. A Phase 1 Randomized Dose-Escalation Study of a Human Monoclonal Antibody to IL-6 in CKD. Kidney360. 2020 Dec 4;2(2):224-235. doi: 10.34067/KID.0005862020. eCollection 2021 Feb 25. PMID 35373026